CLINICAL TRIAL: NCT07338409
Title: Evaluation of Postoperative Outcomes and Mortality in Laparoscopic and Robotic Distal Pancreatectomy: a Retrospective Single-center Analysis
Brief Title: Evaluation of Postoperative Outcomes and Mortality in Laparoscopic and Robotic Distal Pancreatectomy
Acronym: PREINSTRUCT
Status: Completed | Type: Observational
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Dr, PhD, Jessa Hospital
Other Study IDs: 2025/109
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Distal Pancreatectomy (DP)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Minimally invasive distal pancreatectomy can be performed using either a laparoscopic or robotic approach. These minimally invasive techniques are becoming increasingly common in the surgical treatment of both benign and malignant pancreatic lesions. They offer several advantages over traditional open surgery, such as less postoperative pain, better cosmetic results, faster recovery, less blood loss during surgery, and lower healthcare costs. However, despite these advantages, evidence comparing postoperative outcomes, particularly complications, between laparoscopic and robotic distal pancreatectomy remains limited.

Previous studies suggest that robotic surgery may offer technical benefits, such as greater accuracy and precision, which could potentially result in fewer complications. However, the available literature is diverse and often based on small cohorts.

DETAILED DESCRIPTION:
Aim The aim of this study is to evaluate and compare the occurrence and severity of postoperative complications in the 90-day post-operative period between patients undergoing laparoscopic and robotic distal pancreatectomy.

Design A single center retrospective cohort study analysis of patients that underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 30/06/2025.

Sample size All patients that underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 30/06/2025 were included in the study. This were 103 patients.

Study population

Inclusion and exclusion criteria:

All patients that underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 30/06/2025

Primary outcome To to evaluate and compare the occurrence and severity of postoperative complications in the 90-day post-operative period between patients undergoing laparoscopic and robotic distal pancreatectomy.

Secondary outcome measurements Secondary outcome measurements include the evaluation of the Comprehensive Complication Index (CCI), the conversion rates, length of hospital stays, readmission rates, mortality, and the number of lymph nodes harvested. Potential differences in medical costs will also be assessed.

Statistical analysis All data will be transferred from the platform into SPSS Version 28. For descriptive purposes, continuous data are shown as mean ± standard deviation (SD) or median (IQR) for nonnormally distributed data, and categorical data are presented as frequencies (%). For comparative analyses, the Chi-square or Fisher's exact test will be used for categorial variables, and the Independent t-test or Mann-Whitney U test for continuous variables. To assess the primary objective, a bivariate logistic regression model will be used. A P-value <0.05 was considered statistically significant.

Additional collected parameters that are not part of the mandatory registration for complex pancreatic surgery in Belgium are listed below:

- All relevant direct medical costs (e.g., consultation fees and medication) that arise from inpatient care provision will be collected using the financial records of the Jessa Hospital

Additional collected parameters are listed below and are collected as part of the mandatory registration for complex pancreatic surgery in Belgium in the Belgian Cancer Registry (BCR), specifically the "Complex Pancreatic Surgery" registration module:

* Administrative and demographic data
* Referral
* Clinical indication and diagnosis
* Diagnostic procedures
* Comorbidities
* Use of antithrombotic medication
* Neoadjuvant treatment
* Surgery details
* Postoperative outcomes
* Adjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* Underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 31/12/2024.

Exclusion Criteria:

* Underwent open procedure
* Restpancreatectomy
* Central pancreatectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients that underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 31/12/2024 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
90-day postoperative complications | 90- days postoperative
  Postoperative in-hospital complications in the 90-day postoperative period

SECONDARY OUTCOMES:
Cumulative postoperative morbidity | Patients that underwent distal pancreatectomy surgery at Jessa Hospital from 01/01/2020 up until 30/06/2025
  Cumulative postoperative morbidity, quantified using the Comprehensive Complication Index (CCI), which integrates all complications weighted by severity
Length of hospital stay | Time between start of surgery and discharge of hospital
  Length of stay (days) starting from the moment of surgery
Re-admissions | within 30 days of discharge
  Re-admission within 30 days of discharge (from the center that performed the surgery)
Conversion rate | Time from surgery until last follow up of the study
  The rate at which planned minimally invasive surgeries (laparoscopic/robotic) are converted to open surgeries
Mortality | Until the end of the study (31/12/2025)
  Mortality up until 31/12/2025
Lymph nodes harvested | During surgery
  The number of lymph nodes that were retrieved during surgery
Medical costs | From surgery until end of the study (31/12/2025)
  Potential differences in medical costs will be assessed by means of a health-economic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No